CLINICAL TRIAL: NCT01588964
Title: Surgery and Intraperitoneal Hyperthermic Chemotherapy in Patients With Platinum Sensitive Recurrent Ovarian Cancer .
Brief Title: IPHC in Patients With Platinum-sensitive Recurrent Ovarian Cancer
Acronym: IPHC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Clinical Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prot.lf.P.177(A.200)/C.E./2005
Record Dates: First submitted 2012-04-24; First posted 2012-05-01 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Ovarian Epithelial Cancer Recurrent
Keywords: HIPEC; ovarian cancer; recurrence
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIPEC (Experimental): Surgery plus HIPEC
  Interventions: Procedure: HIPEC

INTERVENTIONS:
Procedure: HIPEC — surgery plus HIPEC with the closed technique(perfusion of the abdominal cavity with a solution containing oxaliplatin 460 mg/m2 in 2L/m2 heated saline at 42°C).The global temperature will be measured by thermometer inserted into the esophagus and rectum. A Swan-Ganz catheter will be kept in place during the HIPEC for monitoring cardiovascular function.
  Other Names: IPHC; Hypertermic intraperitoneal chemotherapy

SUMMARY:
In patient with a platinum sensitive ovarian cancer recurrence is demonstrated that the re-challenge with a compound of platinum-based, or a treatment with carboplatin in combination with paclitaxel , determines a rate of clinical response similar to the primary treatment, which is all the more important as the longer the time to progression from the primary therapy.In the clinical setting there are many studies that have shown activity of oxaliplatin and docetaxel in patients with advanced ovarian cancer. Two recent studies have shown clinical efficacy of the combination carboplatin / docetaxel in the first line oxaliplatin / paclitaxel to recurrence of disease, confirming the data already obtained from studies of activity in a single agent.In surgery it has been demonstrated in a meta-analysis including approximately 7000 patients in advanced stages of disease, that the extent of cytoreduction is the most powerful determinant of survival.The role of secondary surgical cytoreduction in case of recurrent disease has yet to be determined because of the lack of prospective randomized clinical studies that may highlight the superiority of such aggressive treatment.The combination of aggressive cytoreductive surgery and hyperthermic intraperitoneal intraoperative chemotherapy (CHIP) used in recent clinical studies showed a prolonged time to progression and disease-free survival in patients with ovarian cancer. However, these studies were conducted on groups of patients with very different among themselves and with other drugs, it is difficult to draw definitive conclusions.Given the activities of oxaliplatin and docetaxel and their non-cross-resistance we designed a Phase 2 clinical trial on treatment of patients with recurrent ovarian cancer, platinum-sensitive, treated with surgical cytoreduction with hyperthermic oxaliplatin-based intraoperative intraperitoneal chemotherapy and following consolidation treatment with oxaliplatin and docetaxel systemically every 21 days.

DETAILED DESCRIPTION:
Among the malignancies of the female genital tract, ovarian cancer is the second most common cancer after the endometrial tumor, but the more lethal, representing the fifth leading cause of death among women in industrialized countries. For the most part, these are epithelial tumors (>70%), who begin with vague gastrointestinal symptoms, general malaise, abdominal bloating, weight loss and fatigue. Because of the non-specificity oh the symptoms and the often late presentation, about 70% of the diagnosis is made at an advanced stage of disease (IIIC). In the last two decades only a modest improvement in survival was achieved. Moreover, even after optimal cytoreduction followed by adjuvant chemotherapy based on platinum and taxane, which is currently the standard for this type of disease, most patients with stage III disease developed a recurrence.

Rational of HIPEC in recurrent ovarian cancer: the cytoreduction. Contrary to what happens in the primary disease is not yet clear what is the standard treatment in recurrent epithelial ovarian cancer (EOC).

Patients who experience a recurrence within 6 months from the end of the first-line chemotherapy are considered platinum-resistant and have applied for a salvage treatment with second line drugs with low response rates and poor survival. Patients who recur after 6 months are considered platinum-sensitive and, therefore, subject to a new chemotherapy treatment with a platinum compound possibly in combination with paclitaxel (re-challenge). In these patients it is possible to achieve a clinical response rate similar to the primary treatment, with median survival reported between 12 and 24 months. Recently surgery affirmed a major role not only in the primary treatment but also in recurrent chemo-sensitive ovarian cancer. A meta-analysis of 2019 patients has shown that obtain an optimal secondary cytoreduction independently correlates with survival (OS) after recurrence. However, a recent Cochrane, showed that, from the studies available nowadays, is not possible to substantiate a difference in prognosis between the exclusive chemotherapy treatment and the association of surgery with adjuvant chemotherapy.

The results of the multicenter trial DESKTOP I show that, even in the presence of peritoneal carcinomatosis, the 2-year survival improves if an optimal cytoreduction is obtained.

Rational of HIPEC in recurrent ovarian cancer: intraperitoneal chemotherapy Many patients who undergo optimal cytoreduction may benefit from adjuvant chemotherapy administered intraperitoneally (IP). Several randomized trials have demonstrated improved survival associated with IP platinum-based chemotherapy as first-line adjuvant therapy after optimal cytoreduction, although it is still unclear which patients might benefit most, or what would be the best drug , its dose or the right number of cycles. The adjuvant IP therapy, however, seems to have more side effects than intravenous therapy (IV) and consequently a worsening of the quality of life (QOL).

Rational use of HIPEC in recurrent ovarian cancer: hyperthermia The association of hyperthermia plus chemotherapy to the surgery based its rational on the cytotoxic effect of hyperthermia, which not only cause a rupture of cell membranes due to protein denaturation (direct effect), but also an increase in the permeability of new vessels and an impairment of receptor protein complexes (indirect effect). The sensitivity of the solid tumors to hyperthermia is probably linked to the creation of a microenvironment with a low pH, low oxygen tension, low glucose levels in response to high temperature. Inactivation of tumor cells is time and temperature dependent, and starts at 40-41 ° C. Experimental data show that human tumor cell lines are more sensitive to a moderate hyperthermia (41-42 ° C).

Furthermore, the ability of its cytotoxic chemotherapeutic agents, including mitomycin C, doxorubicin, cisplatin and oxaliplatin, is enhanced by hyperthermia itself.

Secondary cytoreduction (CRS), HIPEC and ovarian cancer Since its first appearance in 1980, the HIPEC associated with surgery has had an increasingly important role in the treatment of several types of cancer with peritoneal dissemination.

The rational for this therapeutic approach is based on the achievement of higher drug concentrations in contact with the peritoneal surface with a lower systemic concentrations, resulting in a decrease in the systemic toxicity of treatment. The addition of hyperthermia proved to be able to have a cytotoxic effect on tumor cells directly and indirectly, and a synergistic effect with several cytotoxic agents.

Two recent trials including heterogeneous populations of patients with EOC have demonstrated that the use of the HIPEC in association with CRS is followed by an overall survival (OS) of three years after the recurrence that vary between 20-63%. Data from a trial which took place at this Institution and was recently published about the use of HIPEC platinum-sensitive recurrent EOC patients, showed a median disease-free interval (PFS) and OS of 24 and 38 months respectively, with an estimated PFS and OS at 3 years of 44% and 92% respectively. These data not only confirm those previously reported in the literature, but are more significant, probably because of the highly selected population, a characteristic that contrasts with the wide heterogeneity of most of the other trials made until now.

In fact, as demonstrated by the meta-analysis by Bristow et al, the median survival after recurrence in the same group of patients treated with CRS and standard adjuvant chemotherapy alone was 30.3 months. This difference in survival compared with that of our trial could be justified by the increased rate of optimal cytoreduction obtained in our Institution (95.3% vs. 52.2%).

In addition, on the basis of the criteria developed by Markman, that any second-line treatment after recurrence which reaches a PFS similar or comparable to that after the primary disease is considered to be effective, our data show an additional benefit obtained by HIPEC. In the series of patients underwent CRS + HIPEC at this Institution, in fact, the median PFS after primary disease was substantially equal to that after recurrence with values of 25 and 24 months respectively (p = ns). Therefore treatment with CRS associated with HIPEC in with platinum-sensitive recurrent EOC patients would seem to offer the same opportunities in terms of prognosis than primary treatment.

Regarding the complications linked to this procedure, the trials completed at our Institution, showed morbidity and mortality rates about of 35% and 0%, consistent with the data presented by recent review (12 - 52% and 0,9-5,8% respectively), which are however more heterogeneous due to differences between the considered studies. In addition, the analysis divided into two blocks per year of execution of the procedure, has demonstrated a significant reduction in the percentage of complications (up to 26.7%) with a statistically significant difference.

Currently, despite the presence of a strong biological and pharmacological rational and the over 10 years application in EOC, the use of HIPEC in the clinical practice continues to receive mixed reviews. The limit to the confidence in this procedure is the lack of randomized clinical trials and the heterogeneity of the different phase II studies conducted, which resulted in a lack of scientific evidence level I-II. Moreover, the finding of high rates of the related morbidity and mortality, has precluded the use of this procedure to many patients with peritoneal disease.

The primary objective of this trial is therefore to assess whether the use of CRS in combination with HIPEC is able to offer an effectively advantage in terms of survival compared to the exclusive optimal CRS or the only chemotherapy, in platinum-sensitive recurrent EOC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 and under 70 years
* Patients affected by a first recurrence of ovarian cancer with measurable lesions or not, but evaluable (upwards of Ca125 for 2 consecutive assessments).
* ECOG-performance status ≤ 2
* Ovarian cancer limited to the abdominal cavity with or without extraperitoneal spread considered resectable at intraoperative evaluation
* Evidence of tumor recurrence diagnosed after 6 months from primary treatment
* Previous-based chemotherapy of carboplatin and taxanes
* Positive Peritoneal Washing in the presence of other abdominal disease surgically resectable
* Adequate respiratory, hepatic, cardiac, kidney and bone marrow function (absolute neutrophil count > 1500/mm3, platelets > 150,000/μl, creatinine clearance > 60 mL/min according to Cockroft formula)
* Patient-compliant and psychologically able to follow the trial procedures

Exclusion Criteria:

* Non-epithelial ovarian cancer or borderline ovarian tumor
* Pregnancy or breastfeeding
* Patients affected by major depressive disorder even in treatment or minor mood disorders
* Patients with severe impairment of respiratory, hepatic or renal function
* Patients with cardiac, neurological or metabolic uncontrolled pharmacologically disease
* Patients with active infection or other neoplastic disease in progress
* Patients with bowel obstruction
* Inadequate bone marrow, liver, kidney function
* No clear-peritoneal disease at surgical exploration
* Patients with ascites > 500 ml (the TAC)
* Patients on maintenance therapy with Antiangiogenic drugs
* Patients with secondary or tertiary recurrence, or already submitted to HIPEC
* Patients who have already made the second or third line chemotherapy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-03; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival,Overall survival, post operative complications(bowel obstruction,intestinal perforation, hemathologic toxicity (granulocytopenia,thrombocytopenia,anemia),neuropathy. | 6-32 months
  Efficacy and tolerability of the treatment with intraoperative intraperitoneal hyperthermic chemotherapy with oxaliplatin after optimal debulking surgery in patients with platinum-sensitive recurrent ovarian cancer followed by systemic chemotherapy with docetaxel 75mg / m g1 and oxaliplatin 100 mg / m² every 21 days x g1 for six consecutive cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Fagotti, MD, PhD, Principal Investigator — Catholic University of Sacred Heart; Gabriella Ferrandina, MD, Principal Investigator — Catholic University of Sacred Heart; Ida Paris, MD, Principal Investigator — Catholic University of Sacred Heart

REFERENCES:
- [Derived] Fagotti A, Petrillo M, Costantini B, Fanfani F, Gallotta V, Chiantera V, Turco LC, Bottoni C, Scambia G. Minimally invasive secondary cytoreduction plus HIPEC for recurrent ovarian cancer: a case series. Gynecol Oncol. 2014 Feb;132(2):303-6. doi: 10.1016/j.ygyno.2013.12.028. Epub 2013 Dec 27. PMID 24378877